CLINICAL TRIAL: NCT01396122
Title: A Prospective, Multicenter Study to Evaluate the Clinical Performance of the GYNECARE PROSIMA* Pelvic Floor Repair System as a Procedure for Symptomatic POP-Q Stage II-III Pelvic Organ Prolapse
Brief Title: Clinical Performance of GYNECARE PROSIMA* Pelvic Floor Repair System for Symptomatic Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-gyn-02
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2011-07

CONDITIONS: Pelvic Organ Prolapse; Stage II-III
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PROSIMA group (Experimental): Reconstructive surgeries with GYNECARE PROSIMA* were performed in all patients.
  Interventions: Procedure: Procedure: GYNECARE PROSIMA* Pelvic Floor Repair System

INTERVENTIONS:
Procedure: Procedure: GYNECARE PROSIMA* Pelvic Floor Repair System — Perform surgery with GYNECARE PROSIMA* Pelvic Floor Repair System. Vaginal hysterectomy or mid-urethral sling procedure for incontinence could be performed concurrently.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the GYNECARE PROSIMA* Pelvic Floor Repair System as a Device in Women with Symptomatic Pelvic Organ Prolapse.

DETAILED DESCRIPTION:
The GYNECARE PROSIMA* system is a new technique and now available in China. It provides a simplified unanchored mesh repair, making surgery much simpler to perform and reduces the risk of the specific complications that may occur when tunneling devices beyond the pelvic cavity.

In clinical practice, many women have symptomatic prolapse, which requires surgical correction. They are relatively young, and therefore care more about the long-term outcomes and quality of life after procedure. The purpose of this multicenter and prospective study is to evaluate the effectiveness and safety of the GYNECARE PROSIMA* system in the treatment of symptomatic POP-Q Stage II-III pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic pelvic organ prolapse of ICS POP-Q Stage II or III, suitable for surgical repair. Vaginal hysterectomy and mid-urethral sling procedures for incontinence may be performed concurrently.
* Age ≥ 18 years.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires, and documents this agreement by signing the Ethics Committee approved informed consent.

Exclusion Criteria:

* Additional surgical intervention concurrent to the procedure (e.g. sacrocolpopexy, paravaginal repair, tubal sterilisation).
* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Previous hysterectomy within 6 months of scheduled surgery.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* Chronic cough not well-controlled.
* BMI≥30.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Anatomical improvement according to POP-Q score. | 4 weeks
Anatomical improvement according to POP-Q score. | 6 months
Anatomical improvement according to POP-Q score. | 12 months
Anatomical improvement according to POP-Q score. | 2 years
Anatomical improvement according to POP-Q score. | 3 years

SECONDARY OUTCOMES:
Hospital data including operative time, estimated blood loss, length of stay, maximum temperature, time of voiding recovery. | At discharge, an expected average of 5 days after operation.
Pain score measured using Visual Analog Scale (VAS). | 24 hours after surgery and postoperation visit at the 3-4 weeks.
Discomfort of balloon removal, measured using VAS at time of removal. | 24 hours after surgery.
Subject discomfort of VSD by VAS. | postoperation visit at 3-4 weeks.
Presence/absence of complications (composite score) | Up to 6 weeks.
  The occurrence (in the per-operative phase or within 6 weeks post-op) of at least one of the following: 1) bleeding complications; 2) infectious complications; 3) any wound caused by a surgeon movement: bladder, ureteral, or vascular injuries; 4)medical complications: deep vein thrombosis, pulmonary embolism and etc. Complications will be categorized using the Dindo surgical complication grading scale.
Change from baseline in PFIQ-7 scores. | 6 months, 12 months, 2 years and 3 years.
In subjects sexually active at baseline, assessment of sexual function using PISQ-12 (mean scores and change from baseline). | 6 months, 12 months, 2 years and 3 years.
Subject global impression assessed on a 5 point Likert scale. | 6 months, 12 months, 2 years and 3 years.
Presence/absence of complications (composite score) | Up to 3 years.
  Long-term negative outcomes of the surgical procedure will also be recorded until 3 years after surgery. For example, mesh erosion, de novo urinary incontinence, de novo dyspareunia and overall failure rate. Complications will be categorized using the Dindo surgical complication grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (25):
- China (25):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xiamen First Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The First Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The People's Hospital of Hubei Provincial, Wuhan, Hubei
  - The Third Hospital of Wuhan, Wuhan, Hubei
  - The Second Hospital of Xiangya,Central South University, Changsha, Hunan
  - The First Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Maternal and Child Health Hospital, Nanjing Medical University, Wuxi, Jiangsu
  - Affiliated Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital, Shandong University, Jinan, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Fifth People' Hospital of Chengdu, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Beijing Chaoyang Hospital Affiliated to Capital University of Medical Sciences, Beijing
  - The First Affiliated Hospital of Chinese PLA General Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Chongqing Medical University, Chongqin